CLINICAL TRIAL: NCT00176501
Title: Immunotherapy for Patients With Renal Cell Carcinoma
Brief Title: Irradiated Donor Lymphocytes in Treating Patients With Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000540187; P30CA072720 (NIH); CINJ #080410 (Other: CINJ)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-11

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; clear cell renal cell carcinoma; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irradiated allogeneic lymphocytes (Experimental)
  Interventions: Biological: therapeutic allogeneic lymphocytes

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes — If a partially HLA-matched donor is identified and other eligibility criteria are met, the patient will receive irradiated lymphocyte infusion(s).

SUMMARY:
RATIONALE: When irradiated donor lymphocytes are infused into the patient they may help the patient's immune system kill tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving irradiated donor lymphocytes works in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with metastatic renal cell carcinoma treated with HLA-partially matched related donor lymphocytes.
* Determine the rate and kinetics of clinical/radiological response in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the rates of graft-vs-host disease in patients treated with this regimen.

OUTLINE: Patients receive irradiated donor lymphocytes IV over 1 hour on day 0. Treatment repeats every 8-16 weeks for up to 6 donor lymphocyte infusions in the absence of disease progression or unacceptable toxicity.

Blood is collected periodically for research studies, including immunophenotypic analysis of cells and assay for cytotoxic T-lymphocytes and natural killer-cell activity against target cells.

After completion of study treatment, patients are followed for 60 days.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of clear cell renal cell carcinoma

  * Metastatic disease
* Measurable disease
* Previously treated with high-dose aldesleukin OR not eligible for or refused such therapy
* No brain metastases by MRI or CT scan
* HLA-partially matched (e.g., ≥ 2/6 HLA A, B, Dr match) related donor available

  * Patients who have no partially matched immediate family member available are eligible if they have a fully HLA-matched donor

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Bilirubin ≤ 2 times upper limit of normal
* Creatinine clearance ≥ 40 mL/min
* AST ≤ 3 times ULN
* Cardiac ejection fraction ≥ 45%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three subjects were enrolled from March 2005 through February 2006 at Rutgers Cancer Institute of New Jersey, a comprehensive cancer center.
Groups:
- Irradiated Allogeneic Lymphocytes: therapeutic allogeneic lymphocytes : If a partially HLA-matched donor is identified and other eligibility criteria are met, the patient will receive irradiated lymphocyte infusion(s).
Period: Overall Study
Arm/Group | Irradiated Allogeneic Lymphocytes
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Irradiated Allogeneic Lymphocytes
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 55.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: With regard to responses, this trial will use a two-stage Simon's design optimized to minimize the expected number of patients accrued into the study. The maximum sample size will be 35 subjects. 18 subjects will be accrued during stage 1. If there are 2 or fewer responses during this stage, the trial will be stopped early. If there are 3 or more responses during this stage, an additional 19 patients will be accrued for stage 2. If 6 or fewer responses (out of 35) are observed by the end of the trial, then no further investigation of this therapy is warranted.
Time Frame: 5 years
Population: The study was closed early due to slow accrual and insufficient data were collected to analyse this outcome measure.
Arm/Group | Irradiated Allogeneic Lymphocytes
Number analyzed (Participants) | 0

2. Secondary Outcome: Rate and Kinetics of Clinical/Radiological Response
Time Frame: 5 years
Population: The study was closed early due to slow accrual and insufficient data were collected to analyse this outcome measure.
Arm/Group | Irradiated Allogeneic Lymphocytes
Number analyzed (Participants) | 0

3. Secondary Outcome: Rate of Graft-vs-host Disease
Time Frame: 5 years
Population: The study was closed early due to slow accrual and insufficient data were collected to analyse this outcome measure.
Arm/Group | Irradiated Allogeneic Lymphocytes
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Irradiated Allogeneic Lymphocytes
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irradiated Allogeneic Lymphocytes (N=3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Positive lymphocyte culture (Blood and lymphatic system disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irradiated Allogeneic Lymphocytes (N=3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Alkaline phosphatase (Investigations) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Blood and lymphatic system disorders) | 1 (2)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Blood and lymphatic system disorders) | 1 (1)
Pain - Back (General disorders) | 1 (1)
Pain - Kidney (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes